CLINICAL TRIAL: NCT06058078
Title: A Multicenter Phase I/II Clinical Trial to Evaluate the Safety, Tolerability, and Efficacy of RY_SW01cell Injection Therapy in Active Lupus Nephritis
Brief Title: RY_SW01 Cell Injection Therapy in Active Lupus Nephritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Renocell Biotech Company (Industry)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Sun Lingyun, MD, Professor, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RYSW202201
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Lupus Nephritis
Keywords: RY_SW01 cell injection
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RY_SW01 group 1 does 1 RY_SW01 cell injection (Experimental): Receive the best basic treatment and one million cells per kilogram of body weight
  Interventions: Drug: RY_SW01 cell injection; Drug: Basic treatment
- RY_SW01 group 2 does 2 RY_SW01 cell injection (Experimental): Receive the best basic treatment and two million cells per kilogram of body weight
  Interventions: Drug: RY_SW01 cell injection; Drug: Basic treatment
- control group (Other): Receive the best basic treatment
  Interventions: Drug: Basic treatment

INTERVENTIONS:
Drug: RY_SW01 cell injection — Injected RY_SW01 allogonic umbilical cord-derived mesenchymal stem cells(UCMSCs)
  Other Names: UC-MSC treatment
  Arms: RY_SW01 group 1 does 1 RY_SW01 cell injection; RY_SW01 group 2 does 2 RY_SW01 cell injection
Drug: Basic treatment — Drugs for LN treatment
  Other Names: Immunosuppressive drugs

SUMMARY:
RY_SW01 Cell Injection's preclinical research results have shown that the injection significantly improved urine biochemical indicators and tissue damage in two lupus nephritis animal models after MSC administration, with no occurrence of rejection and excellent safety. The mechanism of action of RY_SW01 Cell Injection is relatively clear, demonstrating favorable therapeutic effects in preclinical animal models. Compared to existing conventional therapies, it has the advantages of "convenient treatment and sustained efficacy." It may help reduce the variety and quantity of drugs administered to patients and the various side effects associated with drug treatment. In some cases, it may even lead to the discontinuation of immunosuppressive drugs, reducing mortality and disability rates while improving the quality of life for patients. Its unique advantages have the potential to fundamentally change the current clinical treatment landscape and offer promising prospects for clinical application.

DETAILED DESCRIPTION:
This trial is an exploratory study, including two stages: the dose-escalation phase (Phase I) and the dose-expansion phase (Phase II), as part of a multicenter clinical trial. The Phase I dose-escalation stage employs a dose-escalation trial design, aiming to evaluate the safety, tolerability, and preliminary efficacy of RY_SW01 cell injection in treating patients with active lupus nephritis.

The Phase II dose-expansion stage utilizes a randomized controlled trial design to further evaluate the safety and effectiveness of RY_SW01 cell injection.

The baseline treatment in this trial includes steroids in combination with immunosuppressants. Common immunosuppressants include mycophenolate mofetil, mycophenolate sodium, cyclophosphamide, azathioprine, and calcineurin inhibitors (cyclosporine or tacrolimus), which will be chosen by the researchers based on the patient's condition. During Phase II, the subject's existing baseline treatment regimen must not be increased or changed. If a subject's treatment is assessed as ineffective or intolerable and continuing the existing baseline treatment regimen will not yield better benefits, they may withdraw from the trial and then change their treatment plan or increase the dosage. Such subjects should be included in the effectiveness analysis.The trial will enroll active lupus nephritis patients aged ≥18 and ≤65 years, who must meet all inclusion criteria and none of the exclusion criteria.

Approximately 69-78 subjects are planned to be enrolled to undergo the dose-escalation and dose-expansion trials with RY_SW01 cell injection. About 9-18 evaluable subjects will be enrolled in the dose-escalation stage, and approximately 60 subjects in the dose-expansion stage.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign an informed consent form.
2. Male or female aged ≥18 and ≤65 years.
3. Medical history indicating the fulfillment of at least 4 out of the 11 SLE classification criteria recommended by the American College of Rheumatology (ACR) in 1997, with a Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) score of ≥6.
4. Previous receipt of induction therapy (combination of steroids with immunosuppressants, biologics, or two or more treatments), as determined by the investigator, and the participant demonstrated intolerance to or lack of response to this treatment.
5. Confirmed diagnosis of class III or class IV lupus nephritis according to the ISN/RPS classification criteria (Class III(A), Class III(A+C), Class IV(A), or Class IV(A+C)), with the possibility of being combined with Class V or isolated Class V (including activity and chronicity indices).
6. Laboratory examination showing a urinary protein-to-creatinine ratio (UPCR) > 1000 mg/g or 100 mg/mmol or > 1.0.
7. During the trial and for at least 1 year after injection administration, the participant has no plans for pregnancy and voluntarily agrees to use effective contraception with their partner (see Appendix 1) and has no plans for sperm or egg donation.

Exclusion Criteria:

1. Severe liver dysfunction with any of the following abnormalities: total bilirubin > 2 times the upper limit of normal (ULN); ALT or AST > 2 times the ULN.
2. Severe kidney dysfunction with eGFR < 30 mL/min/1.73m² or serum creatinine > 265.2 µmol/L.
3. Kidney biopsy pathology indicating ≥50% glomerulosclerosis.
4. Blood system abnormalities with any of the following abnormalities: white blood cell count < 2000/µL (2×10^9/L), hemoglobin < 6g/dL (60g/L), platelet count < 30000/µL (30×10^9/L), neutrophils < 1000/µL (1×10^9/L).
5. Severe and uncontrolled cardiovascular diseases, neurological disorders, pulmonary diseases (including obstructive lung disease and interstitial lung disease), liver diseases, endocrine disorders (including uncontrolled diabetes), and gastrointestinal diseases, including but not limited to:

   * Patients with uncontrolled severe hypertension (≥160/100 mmHg).
   * Patients with uncorrected heart failure or severe heart dysfunction (NYHA class ≥III).
   * Patients with a history of myocardial infarction within the previous 6 months or meet the diagnostic criteria for acute myocardial infarction at screening.
   * Patients with a history of acute stroke within the previous 6 months or at risk of acute cerebrovascular events at screening.
   * Patients with a history of severe pulmonary hypertension.
   * Patients with severe arrhythmias (e.g., rapid atrial fibrillation, atrial flutter, paroxysmal ventricular tachycardia).
6. Patients with a history of IgA deficiency (IgA < 10 mg/dL).
7. Patients with other autoimmune diseases except for SLE, including dermatomyositis/polymyositis, mixed connective tissue disease, systemic sclerosis, rheumatoid arthritis, etc., should be excluded. However, patients with secondary Sjögren's syndrome are allowed to participate in this trial.
8. Received live vaccines or attenuated live vaccines within the previous 12 weeks or expect to receive/require live vaccines during the trial.
9. Underwent plasmapheresis or immunoadsorption therapy within the previous 24 weeks or received intravenous immunoglobulin (IVIG) therapy within the previous 4 weeks.
10. Used other investigational drugs within the previous 12 weeks.
11. Tested positive for human immunodeficiency virus antibodies (anti-HIV-Ab) during screening, active syphilis, active hepatitis C (positive for hepatitis C antibodies, and HCV-RNA higher than the lower limit of detection), or positive for hepatitis B surface antigen (HBsAg) and hepatitis B virus DNA (HBV-DNA ≥500 IU/ml).

    History of severe active or recurrent bacterial, viral, fungal, parasitic, or other infections during the screening period.
12. History of malignant tumors within the past 5 years, including solid tumors, hematological malignancies, or in situ cancers (except for surgically removed or cured basal cell carcinoma of the skin).
13. Underwent any major surgery within the previous 12 weeks or anticipated to undergo major surgery during the trial, which is considered to pose an unacceptable risk to the participant by the investigator.
14. Intolerance or contraindication to the treatment protocol of this trial, including any of the following conditions:

    * History of allergies to allogeneic mesenchymal stem cells or excipients (including human albumin).
    * Intolerance or contraindication to oral or intravenous corticosteroids.
    * Absence of peripheral venous access.
15. Pregnant or lactating women.
16. Within the previous 12 months or during the screening period, there is evidence of smoking, alcohol misuse, or drug abuse, defined as follows:

    * Smoking defined as an average daily smoking of ≥5 cigarettes within the previous 3 months.
    * Alcohol misuse defined as consuming more than 14 units of alcohol per week within the previous 3 months (1 unit of alcohol = 350 ml of beer, or 45 ml of spirits, or 150 ml of wine).
    * Drug abuse defined as a positive result in urine drug screening or having a history of drug abuse.
17. Participants judged by the investigator as not suitable for participation in this trial will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events | Within 24 week
Proportion of patients achieving a primary renal efficacy response (PERR) | 24week
Proportion of patients achieving a complete response (CR) | 24week

SECONDARY OUTCOMES:
Frequency of adverse events and severe adverse events | within 24 weeks
Proportion of patients achieving primary renal efficacy response (PERR) | 12 week
Proportion of patients achieving primary renalcomplete response (CR) | 12 week
Changes in urine protein/creatinine ratio (UPCR) relative to baseline | 12 week
Changes in eGFR(estimated glomerular filtration rate)relative to baseline | 12 week
Changes in SLEDAI-2000(The Systemic Lupus Erythematosus Disease Activity Index 2000) ralative to baseline | 24 week
Changes in PGA(Physician Global Assessment) ralative to baseline | 24 week
Changes in SF-36 (Short-form 36 Questionnaire) ralative to baseline | 24 week
The proportion of patients reduced dosage of basic treatment drugs | 24week
Serum biomarkers of antibody | Within 24 weeks
  ANA,nti-dsDNA antibody
the proportion of Treg cell subset | 24 week
Serum biomarkers | Within 24 weeks
  C3,C4
Serum biomarkers of cytokins | Within 24 weeks
  TGF-β，IFN-γ，IL-6,IgG,CXCL10

CONTACTS AND LOCATIONS:
Overall Officials: Sun Lingyun, Principal Investigator — the Affiliated Drum Tower Hospital, Medical School, Nanjing University
Locations (1):
- the Affiliated Drum Tower Hospital, Medical School, Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No